CLINICAL TRIAL: NCT01960400
Title: Investigation of the Efficacy of Transcranial Direct Current Stimulation (tDCS) Added to the Graded Motor Imagery (GMI) in the Treatment of Complex Regional Pain Syndrome (CRPS) Type 1
Brief Title: Investigation of the Efficacy of tDCS in the Treatment of Complex Regional Pain Syndrome (CRPS) Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Yannick Tousignant-Laflamme, PT Ph.D., Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-116
Record Dates: First submitted 2013-09-24; First posted 2013-10-10 (Estimated); Results first posted 2016-11-16 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Reflex Sympathetic Dystrophy
Keywords: Complex regional pain syndrome type 1 (CRPS); Transcranial direct current stimulation (tDCS); Graded motor imagery (GMI); Magnetic resonance imaging (MRI); Functional magnetic resonance imaging (fMRI)
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GMI + tDCS (Active Comparator): Graded motor imagery (GMI) + tDCS
  Interventions: Device: transcranial direct current stimulation (tDCS) (active or placebo); Device: Graded motor imagery (GMI)
- GMI + sham TDCS (Placebo Comparator): Graded motor imagery (GMI) + sham tDCS
  Interventions: Device: transcranial direct current stimulation (tDCS) (active or placebo); Device: Graded motor imagery (GMI)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) (active or placebo) — TDCS was delivered according to the method described by Fregni et al. (2006) and the safety parameters related to tDCS application were respected (DaSilva et al., 2011). Direct current was delivered using a battery-driven constant current stimulator coupled to saline-soaked (0.9% NaCl) sponge electrodes (5 X 7 cm). Anodal stimulation was delivered over the M1; the anode was placed over C3 or C4 position in the 10/20 system for the EEG electrode position, contralateral to the affected limb, and the cathode over the opposite supraorbital area (i.e. ipsilateral to the affected limb). In the laboratory, a constant current of an intensity of 2 mA was applied for 20 min/day X 5 consecutive days during the first and the second weeks of GMI. To help maintain the potential effects of the neurostimulation, the tDCS was also applied simultaneously with GMI once a week during the 2 other phases until the end of the six weeks GMI program, for a total of 14 treatment sessions.
  Other Names: Transcranial direct current stimulation
Device: Graded motor imagery (GMI) — The treatment was performed using a software (Recognise™ online) provided by NOI group (http://www.noigroup.com/recognise). As an alternative to the software (for patients without an internet access), the patient could do the exercises with a Recognise™ Flash Cards set consists of 25 left and 25 right matching images (upper limb or lower limb). Using standardized procedures, inspired from the randomized controlled trial conducted by Moseley (2004, 2006), the participants performed the therapy at home, 10 minutes per session, 3x/day, 6 days/week, using the computer software and a mirror box (Lagueux et al., 2012).

SUMMARY:
The efficacy of the current standard non-pharmacological treatments for complex regional pain syndrome (CRPS), a painful syndrome mostly occurring after musculoskeletal trauma, is suboptimal. It thus appears essential to examine new non-pharmacological therapeutic imagery (GMI) - a non-pharmacological approach with the highest level of evidence (level II). As suggested by the most recent clinical guideline 2, a potential solution would be to add an electrotherapeutic procedure - transcranial direct current stimulation (tDCS) - that may prove effective in modulating cortical excitability and reducing the effect of cortical reorganization on pain. Given the positive results previously obtained in patients with neuropathic pain, it is hypothesized that tDCS will prove to be an innovative add-on treatment method for CRPS patients, and help reduce pain and disability.

DETAILED DESCRIPTION:
Executive summary: The efficacy of the current standard rehabilitation treatments for complex regional pain syndrome (CRPS), a painful syndrome mostly occurring after musculoskeletal trauma, is suboptimal. For instance, the first line of treatment in rehabilitation, progressive motor imagery (GMI), only induces a 50% improvement in symptoms. Although such improvement is interesting, further solutions should be sought to enhance clinical outcomes. It is thus essential to explore new options of therapy. A potential solution to enhance clinical outcomes would be to add an electrotherapeutic procedure, such as transcranial direct current stimulation (tDCS). Given the positive results previously obtained in patients with neuropathic pain, we hypothesize that tDCS will induce functional and structural reorganization in the cortex and lead to better pain relief. The cortical reorganization frequently observed in CRPS patients mainly involves a shrinkage of cortical map of the affected limb on primary and secondary somatosensory cortex. Interestingly, therapies that aim to reverse the cortical reorganization are often associated with a decrease in pain. Therefore, combining GMI and tDCS could lead to added pain relief compared to traditional GMI treatments alone. Furthermore, neuroimaging before and after the procedures could help us explain if and how this is achieved. Objectives: Thus, the primary objective of this research is to study the therapeutic efficacy of tDCS in the treatment of CRPS type 1 in addition to the current best evidence-based rehabilitation treatment, GMI. The second objective is to study, through MRI/fMRI, how brain structures and functions are changed following tDCS and GMI treatments, and whether these changes correlate to clinical changes.

Methodology: To achieve the first objective, we will recruit adults diagnosed with CRPS type 1 via established collaborations with different physicians from our university affiliated hospital. Participants will be randomly allocated into one of the two treatment groups A) experimental group, which will receive the GMI and tDCS stimulation; B) control group, which will receive GMI and sham [placebo] tDCS stimulation. GMI treatment is composed of a three-phase protocol, each lasting two weeks. The GMI treatments will be performed using software and well-established procedures (www.noigroup.com). For its part, the tDCS will be applied for 5 consecutive days during the first 2 weeks of phase 1 and once a week during the 4 other weeks. The anodic (positive) stimulation over the motor cortex (M1) contralateral of the affected limb is sought to modulate cortical excitability and promote pain inhibition and cortical reorganization. Sample size estimates (β:80%,α 5%) show that 15 subjects/group will be necessary.

Anticipated results and impact of the proposed project: This project will allow us to investigate the therapeutic efficacy of an innovative approach to the treatment of CRPS, primarily for the purpose of enhancing the clinical outcomes of GMI. In the event of positive results, we will be able to further examine the therapeutic benefits of this modality in a larger clientele and even in other populations (i.e., patients with chronic low back pain). In addition, our results may contribute to the creation of a clinical practice guide, since there currently is insufficient evidence-based data to establish guidelines regarding the non-pharmacological treatment of CRPS. Finally, MRI/fMRI analysis will help us to capture the phenomenon of tDCS-driven cortical reorganization.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with CRPS type 1, based on Bruehl's diagnostic criteria for research.

Exclusion Criteria:

* Other painful conditions;
* Central nervous system disease;
* Other upper limb conditions;
* Diagnosis of psychiatric condition;
* Dyslexia and/or severe visual impairment;
* Presence of contraindication of tDCS (brain implant, history of severe cranial trauma, severe or frequent headaches, chronic skin conditions);
* Sympathetic blocks for less than one month;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Tousignant-Laflamme, PhD, Principal Investigator — Université de Sherbrooke; Patricia Bourgault, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Sherbrooke, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- GMI + tDCS: Graded motor imagery (GMI) + tDCS
  tDCS: both groups will receive the GMI treatments which will be performed using software and well-established procedures (www.noigroup.com). For its part, the tDCS will be applied for 5 consecutive days during the first 2 weeks of phase 1 and once a week during the 4 other weeks. The anodic (positive) stimulation over the motor cortex (M1) contralateral of the affected limb is sought to modulate cortical excitability and promote pain inhibition and cortical reorganization.
- GMI + Sham TDCS: Graded motor imagery (GMI) + sham tDCS
  tDCS: both groups will receive the GMI treatments which will be performed using software and well-established procedures (www.noigroup.com). For its part, the tDCS will be applied for 5 consecutive days during the first 2 weeks of phase 1 and once a week during the 4 other weeks. The anodic (positive) stimulation over the motor cortex (M1) contralateral of the affected limb is sought to modulate cortical excitability and promote pain inhibition and cortical reorganization.
Period: Overall Study
Arm/Group | GMI + tDCS | GMI + Sham TDCS
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GMI + tDCS | GMI + Sham TDCS | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.91 (10.76) | 52.83 (12.81) | 46.87 (13.06)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity
Description: The choice of outcome measures was performed in accordance with Initiative on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT) guidelines (Dworkin et al., 2005). All instruments were used before (T0) and after 6 weeks of treatment (T1).
  The primary outcome measure was pain severity as measured with the Brief pain inventory short-form (BPI-sf) (Poundja et al., 2007). The BPI-sf includes four questions on pain levels, where subjects were asked to rate intensity on a scale of 0 (no pain) to 10 (worst possible pain) for: (1) pain at its worst in the last 24 hours; (2) pain at its least in the last 24 hours; (3) pain on average in the last 24 hours; (4) pain right now. The total score ranges from 0 to 40 (sum of the four subscales). The higher the score, the greater the severity of the pain is severe.
Time Frame: Before (T0) and after treatment (6 weeks) (T1)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active tDCS + GMI: tDCS: In the laboratory, a constant current of an intensity of 2 mA (subthreshold intensity) was applied for 20 minutes a day for five consecutive days (Monday to Friday) during the first and the second weeks of GMI (see Fig. 1A). To help maintain the potential effects of the neurostimulation, the tDCS was also applied simultaneously with GMI once a week (Monday) during the 2 other phases until the end of the six weeks GMI program, for a total of 14 treatment sessions.
  tDCS + GMI: In the laboratory, after 8 minutes of tDCS application, patients were asked to perform their GMI treatments with the help of a portable computer. Seated comfortably, the patients had to perform the exercises according to the treatment phase for a period of 10 minutes.
- Placebo tDCS + GMI: tDCS: For the group receiving the placebo tDCS, the electrodes were placed in the same position as for active stimulation using the tDCS stimulator, but with the placebo mode automatically turned off after 30 seconds of stimulation). This type of sham stimulation has been shown to reliably blind subjects (Gandiga et al., 2006).
  tDCS + GMI: In the laboratory, after 8 minutes of tDCS application, patients were asked to perform their GMI treatments with the help of a portable computer. Seated comfortably, the patients had to perform the exercises according to the treatment phase for a period of 10 minutes.
Arm/Group | Active tDCS + GMI | Placebo tDCS + GMI
Number analyzed (Participants) | 11 | 11
units on a scale
  Before treatment (T0) | 22.18 (7.43) | 23.36 (6.19)
  After treatment (T1) | 18.00 (9.20) | 23.82 (5.93)
Statistical Analysis 1: Comparison: Active tDCS + GMI vs Placebo tDCS + GMI; For the severity of pain, the calculations have revealed that only this pain now had an acceptable statistical power, of 77.1% after treatment (T1); Test type: Superiority or Other; p = 0.065, ANOVA — The statistical signifiance level : p<0.05. After treatment (T1) Pain severity p=0.065 Sub-scale: * Present pain p=0.046* * Average pain p=0.381 * Most intense pain p=0.064 * Least intense pain p=0.142; To assess the effectiveness of interventions (inter-group differences), a mixed-model ANOVA (time X group interaction) was used

2. Secondary Outcome: Pain Catastrophizing
Description: The Pain catastrophizing scale (PCS) (Sullivan et al., 1995) was used to evaluate the feelings, thoughts, and emotions related to pain catastrophizing of the patient. The PCS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness.
  * The scores ranging from 0 to 52 points (sum of the tree subscales), with higher scores representing stronger pain catastrophizing (Sullivan et al., 1995).
Time Frame: Before (T0) and after treatment (6 weeks) (T1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS + GMI | Placebo tDCS + GMI
Number analyzed (Participants) | 11 | 11
units on a scale
  Before treatment (T0) | 24.09 (10.98) | 27.64 (10.36)
  After treatment (T1) | 16.64 (10.68) | 25.91 (11.42)
Statistical Analysis 1: Comparison: Active tDCS + GMI vs Placebo tDCS + GMI; Test type: Superiority or Other; p = 0.049, ANOVA — interaction group X time

3. Secondary Outcome: Kinesiophobia
Description: The Tampa Scale of kinesiophobia (TSK) (Kori et al., 1990) was used to assess fear of movement and injury/(re)injury. The TSK questionnaires consist of 17 items. Each item, composed of a statement, is scored by the patient on a 4-point Likert scale of 1 (strongly disagree) to 4 (strongly agree). The total scores range from 17 to 68, with higher scores representing stronger fear-avoidance beliefs (Clark, Kori, Brockel, 1996).
Time Frame: Before (T0) and after treatment (6 weeks) (T1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS + GMI | Placebo tDCS + GMI
Number analyzed (Participants) | 11 | 11
units on a scale
  Before treatment (T0) | 44.09 (8.60) | 42.55 (8.59)
  After treatment (T1) | 40.36 (8.23) | 42.82 (8.27)
Statistical Analysis 1: Comparison: Active tDCS + GMI vs Placebo tDCS + GMI; Test type: Superiority or Other; p = 0.035, ANOVA — interaction group X time

4. Secondary Outcome: State Anxiety
Description: The State-Trait Anxiety Inventory (STAI) was used to assess the state of anxiety at the moment (Spielberg et al., 1983). The total score is obtained by adding the scores for all 20 questions range from 20 to 80; the higher the result is, the higher is the anxiety about an event.
Time Frame: Before (T0) and after treatment (6 weeks) (T1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS + GMI | Placebo tDCS + GMI
Number analyzed (Participants) | 11 | 11
units on a scale
  Before treatment (T0) | 41.91 (14.43) | 41.91 (17.61)
  After treatment (T1) | 35.91 (12.19) | 44.00 (15.38)
Statistical Analysis 1: Comparison: Active tDCS + GMI vs Placebo tDCS + GMI; Test type: Superiority or Other; p = 0.046, ANOVA — interaction group X time

ADVERSE EVENTS:
Time Frame: Adverse events were collected each week of the intervention (six weeks). A questionnaire on adverse effects was done after six weeks of treatment (T1). No follow-up was done after the end of treatment.
Groups:
- GMI + Active tDCS: Graded motor imagery (GMI) + active tDCS
- GMI + Placebo tDCS: Graded motor imagery (GMI) + placebo tDCS
Arm/Group | GMI + Active tDCS | GMI + Placebo tDCS
Serious Adverse Events (participants affected / at risk) | 5/11 | 3/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GMI + Active tDCS (N=11) | GMI + Placebo tDCS (N=11)
Increase pain (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Fasciculation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Light headache (Nervous system disorders) | 3 (3) | 2 (2)
Burning sensation (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes